CLINICAL TRIAL: NCT00005047
Title: MVAC (Methotrexate, Vinblastine, Adriamycin, and Cisplatin) in Organ-Confined Bladder Cancer Based on p53 Status
Brief Title: 4B951, Combination Chemotherapy in Treating Patients With Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual was halted on the basis of the Data and Safety Monitoring Board review of a futility analysis.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067639; LAC-USC-4B951 (Other: USC); SWOG-4B951 (Other: SWOG); NCI-G00-1715 (Other: NCI); NYU-9852 (Other: NYU); CAN-NCIC-BL10 (Other: NCIC-CTG); CCCWFU-88198; U10CA032102 (NIH)
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer
Keywords: stage I bladder cancer; stage II bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Doxorubicin; Methotrexate; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I: M-VAC x 3 (Experimental): Patients with altered (+) p53, reconsented to randomization, randomized to three cycles of MVAC
  Interventions: Drug: cisplatin; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: vinblastine
- Arm II: Observation (No Intervention): Patients with altered (+) p53, reconsented to randomization, randomized to observation
- Arm III: Observation (No Intervention): Patients with unaltered (-) p53
- Arm IV: Observation (No Intervention): Patients with altered (+) p53, patients did not consent to randomization

INTERVENTIONS:
Drug: cisplatin
  Arms: Arm I: M-VAC x 3
Drug: doxorubicin hydrochloride
  Arms: Arm I: M-VAC x 3
Drug: methotrexate
  Arms: Arm I: M-VAC x 3
Drug: vinblastine
  Arms: Arm I: M-VAC x 3

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether combination chemotherapy is more effective than observation alone in treating bladder cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy to see how well it works compared to observation alone in treating patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the recurrence-free and overall survival in patients with transitional cell carcinoma of the bladder with p53 gene alterations treated with methotrexate, vinblastine, doxorubicin, and cisplatin vs observation alone.
* Compare the recurrence-free and overall survival in patients with or without p53 gene alterations treated with observation alone.
* Examine the expression of p53 and other genes, particularly RB, p21, and p16, involved in cell cycle regulation that may be involved in the response to chemotherapy in these patients.
* Correlate p53 mutational gene status with p53 protein expression by immunohistochemistry, outcome (recurrence-free and overall survival), response to chemotherapy, and expression of key molecules in the p53-mediated apoptotic pathway in patients treated with this regimen vs observation alone.

OUTLINE: This is a randomized, multicenter study. Patients are assigned to 1 of 2 treatment groups based on the status of the p53 gene in the bladder tumor.

* Group A (p53 gene alteration, defined by greater than 10% nuclear reactivity): Patients are stratified according to age (under 65 vs 65 and over), stage (P1 vs P2a vs P2b), grade (1 or 2 vs 3 or 4), and p21 status. Patients are randomized to 1 of 2 treatment arms within 10 weeks after radical cystectomy and bilateral pelvic lymphadenectomy and within 2 weeks after registration.

  * Arm I: Within 2 weeks after randomization, patients receive methotrexate IV on days 1, 15, and 22; vinblastine IV on days 2, 15, and 22; and doxorubicin IV and cisplatin IV on day 2. Treatment repeats every 4 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients undergo observation for recurrence but do not receive adjuvant chemotherapy after surgery.

Patients who are eligible for randomization but decline to be randomized undergo observation for recurrence.

* Group B (p53 gene normal, defined by less than 10% nuclear reactivity): Patients undergo observation for recurrence but do not receive adjuvant chemotherapy after surgery.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study within 4.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven organ confined transitional cell carcinoma (TCC) of the bladder

  * Must have undergone radical cystectomy and bilateral pelvic lymphadenectomy with pathologic stage from definitive cystectomy specimen of P1, P2a, or P2b and N0, M0 TCC with or without squamous/glandular differentiation (no adenocarcinoma, squamous cell carcinoma, or small cell carcinoma)

    * Margins must be negative for invasive or in situ TCC
    * In situ TCC in the urethra or ureter(s) allowed provided margins are negative
  * Clinical stage T1, T2a, or T2b based on transurethral resection bladder tumor specimen with P0 or PIS and N0, M0 TCC allowed
  * Incidental pT2a (Gleason score no greater than 7), pT2b (Gleason score no greater than 7), or pT2c (Gleason score no greater than 7) adenocarcinoma of the prostate allowed
* No invasive tumor into ureter(s) or urethra
* Must have potentially curable disease
* Must register within 9 weeks after surgery
* No metastatic disease by physical exam and chest x-ray or CT scan of the chest
* Eligible for randomization if:

  * p53 gene alteration present
  * Randomization occurs within 10 weeks after surgery
  * Those who are randomized to receive (MVAC) methotrexate, vinblastine, doxorubicin, and cisplatin begin MVAC within 12 weeks after cystectomy
  * No metastatic disease by physical exam and chest x-ray or CT scan of the chest
  * No prohibitive medical risk for chemotherapy

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 4,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic

* SGOT or SGPT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal
* Bilirubin normal

Renal

* Creatinine no greater than 1.8 mg/dL OR
* Creatinine clearance at least 50 mL/min
* Blood urea nitrogen normal

Cardiovascular

* No serious arrhythmias
* No congestive heart disease with New York Heart Association class III or IV status
* Randomization group:

  * Ejection fraction must be at least 50% by MUGA scan if there is a clinical concern regarding the patient's cardiac status

Other

* No other malignancy (including synchronous papillary or invasive upper urinary tract malignancy) within the past 5 years except incidental prostate cancer (found at cystectomy), basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* No concurrent advanced medical illness or psychologic disease
* No prohibitive medical risk for chemotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior systemic chemotherapy for bladder cancer
* At least 5 years since other prior systemic chemotherapy
* Prior intravesical therapy allowed
* Randomization group:

  * Prior intravesical therapy allowed if administered prior to cystectomy

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic irradiation

Surgery

* See Disease Characteristics

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 1997-08 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Cote, MD, FRCPath, Study Chair — University of Southern California; Laurence H. Klotz, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Seth P Lerner, MD, Study Chair — Baylor College of Medicine
Locations (74):
- United States (73):
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
- Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] von Rundstedt FC, Mata DA, Groshen S, Stein JP, Skinner DG, Stadler WM, Cote RJ, Kryvenko ON, Godoy G, Lerner SP. Significance of lymphovascular invasion in organ-confined, node-negative urothelial cancer of the bladder: data from the prospective p53-MVAC trial. BJU Int. 2015 Jul;116(1):44-9. doi: 10.1111/bju.12997. Epub 2015 Mar 25. PMID 25413313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with stage pT1/T2N0M0 urothelial cancer who had undergone a radical cystectomy within the prior 9 weeks were eligible for enrollment. Twenty-two patients who were registered were never assigned to a group after enrolling due to: missing baseline documentation (5), incorrect disease stage (13), and patient withdrawal (4).
Groups:
- Arm I: M-VAC x 3: Patients with altered (+) p53, reconsented to randomization, randomized to three cycles of MVAC
  cisplatin
  doxorubicin hydrochloride
  methotrexate
  vinblastine
Period: Overall Study
Arm/Group | Arm I: M-VAC x 3 | Arm II: Observation | Arm III: Observation | Arm IV: Observation
Started | 58 | 56 | 227 | 158
Completed | 39 | 56 | 227 | 158
Not Completed | 19 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: M-VAC x 3: p53 positive, randomized to 3 cycles of adjuvant combination methotrexate, vinblastine, doxorubicin and cisplatin (MVAC)
- Arm II: Observation: p53 positive, randomized to observation/no intervention
- Arm III: Observation: p53 negative, assigned to observation/no intervention
- Arm IV: Observation: p53 positive, refused random assignment, assigned to observation/no intervention
- Total: Total of all reporting groups
Arm/Group | Arm I: M-VAC x 3 | Arm II: Observation | Arm III: Observation | Arm IV: Observation | Total
Number analyzed (Participants) | 58 | 56 | 227 | 158 | 499
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 41 | 127 | 81 | 286
  >=65 years | 21 | 15 | 100 | 77 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 49 | 34 | 99
  Male | 51 | 47 | 178 | 124 | 400
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52 | 49 | 203 | 150 | 454
  Black | 4 | 1 | 13 | 4 | 22
  Asian | 0 | 2 | 6 | 1 | 9
  Hispanic | 1 | 4 | 3 | 3 | 11
  Other | 1 | 0 | 2 | 0 | 3
Stage [Count of Participants; unit: Participants] — The TNM classification for pathologic (p) staging of bladder cancer Primary tumor (T):
  TX Primary tumor cannot be assessed T0 No evidence of primary tumor Ta Noninvasive papillary carcinoma Tis Carcinoma in situ: "flat tumor" T1 Tumor invades subepithelial connective tissue T2 Tumor invades muscularis propria T2a The tumor has spread to the inner half of the muscle of the bladder wall, which may be called the superficial muscle.
  Participants
    pT1 | 21 | 16 | 87 | 61 | 185
    pT2 and pT2a | 37 | 40 | 140 | 97 | 314
Grade [Count of Participants; unit: Participants] — Grade 1: Increased umber of urothelial cell layers, no mitotoc cells identified, slight cytologic atypia Grade 2: Rare mitotic cells identified, mild cytologic atypia with uniform appearing cells Grade 3: Moderate cellular atypia, mitotic cells easily identifiable, variation in cellular appearance Grade 4: Severe cellular atypia, frequent mitotic cells, cellular pleomorphisms, difficult to identify cell of origin
  Participants
    1 or 2 | 2 | 1 | 16 | 5 | 24
    3 or 4 | 56 | 55 | 210 | 152 | 473
    missing | 0 | 0 | 1 | 1 | 2
No. of nodes identified [Count of Participants; unit: Participants]
  <15 nodes | 22 | 14 | 68 | 64 | 168
  >= 15 nodes | 36 | 42 | 159 | 94 | 331
p21 status [Count of Participants; unit: Participants]
  Absent | 24 | 22 | 35 | 64 | 145
  Present | 34 | 34 | 190 | 92 | 350
  missing | 0 | 0 | 2 | 2 | 4
Lymphovascular invasion [Count of Participants; unit: Participants]
  No | 33 | 25 | 117 | 84 | 259
  Yes | 13 | 14 | 46 | 29 | 102
  Unknown | 12 | 17 | 64 | 45 | 138
Bladder carcinoma in situ [Count of Participants; unit: Participants]
  No | 16 | 12 | 60 | 36 | 124
  Yes | 34 | 32 | 137 | 99 | 302
  Unknown | 8 | 12 | 30 | 23 | 73

OUTCOME MEASURES:

1. Primary Outcome: Probability of Recurring
Description: p53 positive patients randomized to MVAC (arm I) compared to p53 positive patients randomized to observation (arm II). Time from registration to the first observation of disease recurrence, censoring patients who died of unrelated causes. Probabilities of recurring were based on cumulative incidence curves.
  Recurrence is defined as first radiological appearance of bladder cancer, per local standard of care.
Time Frame: 5 years
Measure: Median (Standard Error); unit: probability
Arm/Group | Arm I: M-VAC x 3 | Arm II: Observation
Number analyzed (Participants) | 58 | 56
probability | 0.85 (0.05) | 0.84 (0.06)

2. Secondary Outcome: Probability of Overall Survival
Description: p53 positive patients randomized to MVAC (arm I) compared to p53 positive patients randomized to observation (arm II). Survival is calculated from registration to death due to any cause. Probabilities of survival were based on the Kaplan-Meier product-limit method.
Time Frame: 5 years
Measure: Median (Standard Error); unit: probability
Arm/Group | Arm I: M-VAC x 3 | Arm II: Observation
Number analyzed (Participants) | 58 | 56
probability | 0.87 (0.05) | 0.84 (0.05)

3. Secondary Outcome: Probability of Recurrence
Description: Patients with tumors demonstrating alteration in p53 compared to patients with no p53 alterations.
  Probabilities of recurring were based on cumulative incidence curves. Recurrence is defined as first radiological appearance of bladder cancer, per local standard of care.
Time Frame: 5 years
Population: This analysis compares p53 positive patients (combined arms I, II, and IV) to p53 negative patients (arm III).
Measure: Median (Standard Error); unit: probability
Groups:
- p53 Positive Patients: Arm I: Patients with altered (+) p53, reconsented to randomization, randomized to three cycles of MVAC
  Arm II: Patients with altered (+) p53, reconsented to randomization, randomized to observation
  Arm IV: Patients with altered (+) p53, patients did not consent to randomization
- p53 Negative Patients: Arm III: Observation; Patients with unaltered (-) p53
Arm/Group | p53 Positive Patients | p53 Negative Patients
Number analyzed (Participants) | 272 | 227
probability | 0.83 (0.03) | 0.77 (0.03)

4. Secondary Outcome: Probability of Overall Survival
Description: Patients with tumors demonstrating alteration in p53 compared to patients with no p53 alterations. Probabilities of survival were based on the Kaplan-Meier product-limit method.
Time Frame: 5 years
Population: This analysis compares p53 positive patients (combined arms I, II, and IV) to p53 negative patients (arm III).
Measure: Median (Standard Error); unit: probability
Arm/Group | p53 Positive Patients | p53 Negative Patients
Number analyzed (Participants) | 272 | 227
probability | 0.82 (0.03) | 0.84 (0.03)

ADVERSE EVENTS:
Time Frame: 5 years: every 3 months for the first year, every 6 months for the following 4 years
Description: Serious Adverse Events and Other Adverse events were recorded only for Arm I, as all other arms were observation. Adverse events were only recorded for those patients who received MVAC (46/58).
  All-Cause Mortality was monitored for patients in all the Arms.
Arm/Group | Arm I: M-VAC x 3 | Arm II: Observation | Arm III: Observation | Arm IV: Observation
All-Cause Mortality (participants affected / at risk) | 12/58 | 9/56 | 41/227 | 36/158
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 35/46 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: M-VAC x 3 (N=46) | Arm II: Observation (N=0) | Arm III: Observation (N=0) | Arm IV: Observation (N=0)
Decreased WBC (Blood and lymphatic system disorders) | 14 | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 31 | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No